CLINICAL TRIAL: NCT06778824
Title: Esophageal Visceral Hypersensitivity and Hypervigilance in Disorders of Gut-brain Interaction: the Roles of Neuromodulators
Brief Title: Neuroregulators for the Treatment of Diseases Associated With Esophageal-brain-gut Axis Communication Abnormalities.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Lei, Wei-Yi, HualienTCGH, Hualien Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB112-201-A
Record Dates: First submitted 2025-01-05; First posted 2025-01-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Gut-Brain Disorders; GERD Without Erosive Esophagitis
Keywords: gastroesophageal reflux disease; disorders of gut-brain interaction; neuromodulators
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole; Sertraline; Tablets; Imipramine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tricyclic antidepressant, TCA (Experimental): The main component of tricyclic antidepressants (TCA) is imipramine HCL. Imipramine has various pharmacological effects, including alpha-adrenergic antagonism, antihistamine activity, anticholinergic effects, and blockade of 5-HT3 receptors. The exact mechanism of imipramine's antidepressant action is unknown, but it may primarily involve the inhibition of the reuptake of norepinephrine (NA) and serotonin (5-HT), without including a stimulatory effect on the central nervous system.
  Indications/Expected Uses: Depression and nocturia.
  Interventions: Drug: Imipramine Pill
- selective serotonin reuptake inhibitor, SSRI (Experimental): The mechanism of action of the selective serotonin reuptake inhibitor (SSRI) sertraline is believed to be related to the inhibition of serotonin (5-HT) reuptake in the central nervous system. Clinical studies have confirmed that when humans receive appropriate doses of sertraline, it can inhibit the reuptake of serotonin into platelets in the body.
  Indications/Expected Uses: Depression, obsessive-compulsive disorder (OCD), panic disorder, post-traumatic stress disorder (PTSD), social anxiety disorder, and premenstrual dysphoric disorder (PMDD).
  Interventions: Drug: Zoloft 50Mg Tablet
- proton-pump inhibitor, PPI (Experimental): Proton-pump inhibitors (PPIs) inhibit gastric acid secretion by specifically targeting the (H+, K+)-ATPase enzyme system on the surface of gastric parietal cells. This enzyme system can be considered an acid (proton) pump within the parietal cells, blocking the final step of gastric acid production. As a result, they are classified as gastric acid pump inhibitors, effectively reducing both basal and stimulated gastric acid secretion, independent of stimulation. Lansoprazole does not possess anticholinergic or histamine H2-receptor antagonist activity.
  Indications/Expected Uses: Treatment of gastric ulcers, duodenal ulcers, gastroesophageal reflux disease (GERD) with erosive esophagitis, and management of symptoms related to GERD. It is also used in Zollinger-Ellison syndrome, in combination with antibiotic treatment for Helicobacter pylori-related peptic ulcers, and for the treatment of gastric ulcers induced by NSAIDs.
  Interventions: Drug: Takepron

INTERVENTIONS:
Drug: Takepron — Participants are expected to take a proton-pump inhibitor (PPI) for 12 weeks, with a dosage of 30 mg taken once a day.
  Other Names: Takepron ® OD Tablets 15．30mg
  Arms: proton-pump inhibitor, PPI
Drug: Zoloft 50Mg Tablet — Participants are expected to take a selective serotonin reuptake inhibitor (SSRI) for 12 weeks, with a dosage of 50 mg taken once a day.
  Other Names: ZOLOFT Film Coated Tablets 50 mg
  Arms: selective serotonin reuptake inhibitor, SSRI
Drug: Imipramine Pill — Participants are expected to take tricyclic antidepressants (TCA) for 12 weeks, with a dosage of 25 mg taken twice a day.
  Other Names: Tone F.C. Tablets 25mg"MEIDER"(lmipramine hydrochloride)
  Arms: tricyclic antidepressant, TCA

SUMMARY:
Gastroesophageal reflux disease (GERD) poses a challenging medical condition to manage, with up to 40% of patients showing refractory to standard medical intervention, which usually begins with a proton pump inhibitor (PPI). Among these cases, esophageal disorders of gut-brain interaction (DGBI), such as reflux hypersensitivity and functional heartburn, or GERD patients with concurrent occurrences of these conditions, constitute more than 90% of the patients who did not respond to twice-daily PPI treatment. Esophageal visceral hypersensitivity and hypervigilance are the two pathways that drive esophageal DGBI and symptoms. The Rome IV esophageal disorders, encompassing functional chest pain, functional heartburn, globus, functional dysphagia, and reflux hypersensitivity, are defined by present with symptoms originating from the esophagus without detectable evidence of structural, inflammatory, or motor disorders. Diagnosing esophageal DGBI necessitates testing involving endoscopy, pH-impedance monitoring, and high-resolution manometry. Neuromodulators form the basis of the pharmacological strategy for managing various esophageal DGBI and symptoms, modulating both peripheral and central hyperalgesia. Increasing evidence supports the use of brain-gut behavioral therapies, such as gut-directed hypnotherapy and cognitive behavior therapy, as effective treatments for a variety of DGBIs. However, the efficacy of neuromodulators in treating esophageal DGBI and related symptoms remains largely unexplored. The primary objective of this study is to examine the efficacy of neuromodulators in managing esophageal DGBI. Additionally, investigators will explore various classes of neuromodulators and subtypes of esophageal DGBI to ascertain whether there are differing levels of effectiveness across these conditions. The findings from this study will contribute to a better understanding of the pathophysiology of esophageal DGBI and GERD with refractory symptoms. These clinical insights may then offer valuable guidance for future therapeutic approaches in DGBI patients who experience esophageal symptoms and do not respond to PPI treatment.

DETAILED DESCRIPTION:
Procedure steps： n Study One, each participant first completed a questionnaire that included the Gastroesophageal Reflux Disease Questionnaire (GERDQ, PROMIS GERD, DSI & GSS, RSI), the Brief Esophageal Swallowing Difficulty Scale (BEDQ), the Esophageal Hypersensitivity and Anxiety Scale (EHAS), the Visceral Sensitivity Index (VSI), and the Sleep and Psychosocial Questionnaire (Pittsburgh Sleep Quality Index (PSQI), Taiwanese Depression Questionnaire (TDQ), State-Trait Anxiety Inventory (STAI), Functional Dyspepsia (FD) Questionnaire, Irritable Bowel Syndrome (IBS) Questionnaire, and the Quality of Life Questionnaire (SF-12, Northwest Esophageal Quality of Life Scale (NEQOL)). Completing the questionnaires took approximately 20 to 30 minutes.

Afterward, participants were randomly assigned by computer to receive either 12 weeks of treatment with a neuromodulator-tricyclic antidepressants (TCA), or a neuromodulator-selective serotonin reuptake inhibitors (SSRI), or 12 weeks of the control medication-proton pump inhibitors (PPI). Investigators plan to recruit 70 participants for the TCA group, 70 for the SSRI group, and 70 for the PPI group, with each participant having about a 1/3 chance of being assigned to one of these groups.

The tricyclic antidepressant (TCA) will be administered as 25 mg enteric-coated tablets (Department of Health Drug Code 047966), taken twice daily. The selective serotonin reuptake inhibitor (SSRI) will be administered as 50 mg enteric-coated tablets (Department of Health Drug Code 021780), taken once daily. The control medication, the proton pump inhibitor (PPI), will be given as 30 mg orally dissolving tablets (Department of Health Drug Code 024273), taken once daily.

At the end of the 12-week medication treatment, participants will complete another round of questionnaires to conclude the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, with clear consciousness and willingness to sign the informed consent form.
2. Subjects with chronic esophageal symptoms related to disorders of the brain-gut axis communication (such as heartburn, acid reflux, sensation of a foreign body in the throat, difficulty swallowing, and chest pain or discomfort).

Exclusion Criteria:

1. Esophageal strictures, or history of surgery on the esophagus, gastrointestinal tract, or throat.
2. Structural esophageal diseases (such as diverticula, esophageal rings, etc.), infectious esophagitis, erosive esophagitis, eosinophilic esophagitis.
3. Non-erosive gastroesophageal reflux disease or significant esophageal motility disorders.
4. History of or current diagnosis of malignancies in the esophagus, gastrointestinal tract, or other organs.
5. Significant endocrine or rheumatic immune diseases that may affect gastrointestinal motility.
6. Continuous use of medications that may affect esophageal motility within the past month (such as anticholinergics, opioid-like agents, nitrates, calcium channel blockers, etc.).
7. Use of or currently taking antidepressants, selective serotonin reuptake inhibitors, or other psychotropic medications within the past three months.
8. Pregnant or breastfeeding women.
9. Individuals with mental illness or those who are unable to cooperate.
10. Known allergy to tricyclic antidepressants.
11. Known allergy to selective serotonin reuptake inhibitors.
12. Known allergy to any component of proton pump inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal Reflux Disease Questionnaire（GERDQ） | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
PROMIS Gastroesophageal Reflux Disease Questionnaire（PROMIS GERD） | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Disease symptom index(DSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Reflux Symptom Index(RSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
The Brief Esophageal Dysphagia Questionnaire(BEDQ) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Esophageal Hypervigilance and Anxiety Scale(EHAS) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Visceral sensitivity index(VSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Pittsburgh Sleep Quality Index(PSQI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Taiwanese Depression Questionnaire(TDQ) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
The State-Trait Anxiety Inventory(STAI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Functional dyspepsia(FD) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Irritable bowel syndrome questionnaire(IBS) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Short-form-12-health-survey-questionnaire(SF-12) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Northwest Esophageal Quality of Life Scale(NEQOL) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
Global Symptom Severity Questionnaire(GSS) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Gastroenterology attending physician Lei Wei-Yi, Principal Investigator — staff
Locations (1):
- Hualien Tzu Chi Hospital,Buddhist Tzu Chi Medical Foundation, Hualien City, Taiwan

DOCUMENTS (2):
  • Study Protocol (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT06778824/Prot_000.pdf
  • Informed Consent Form (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT06778824/ICF_001.pdf